CLINICAL TRIAL: NCT00621764
Title: A Controlled Study of the Safety and Immunogenicity of ChimeriVax™ Japanese Encephalitis Vaccine in Thai Toddlers and Children
Brief Title: Immunogenicity and Safety of ChimeriVax™ Japanese Encephalitis Vaccine in Thai Toddlers and Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: JEC01
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Japanese Encephalitis; Hepatitis A
Keywords: Japanese encephalitis (JE); Hepatitis A; Inactivated Mouse-Brain
MeSH Terms: conditions — Encephalitis, Japanese; Hepatitis A | interventions — Japanese Encephalitis Vaccines; Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- JE-CV/Hepatitis A (Group 1) (Experimental): Participants aged 2 to 5 years at enrollment; to receive Japanese encephalitis vaccine (Day 0) and Hepatitis A vaccine (Day 28)
  Interventions: Biological: Japanese encephalitis vaccine (Day 0) Hepatitis A vaccine (Day 28)
- Hepatitis A/JE-CV (Group 2) (Experimental): Participants aged 2 to 5 years at enrollment; to receive Hepatitis A vaccine (Day 0) and Japanese encephalitis vaccine (Day 28)
  Interventions: Biological: Hepatitis A vaccine (Day 0) Japanese encephalitis vaccine (Day 28)
- JE-CV/Hepatitis A (Group 3) (Experimental): Participants aged 12 to 24 months at enrollment; to receive Japanese encephalitis vaccine (Day 0) and Hepatitis A vaccine (Day 28)
  Interventions: Biological: Japanese encephalitis vaccine (Day 0) Hepatitis A vaccine (Day 28)
- Hepatitis A/JE-CV (Group 4) (Experimental): Participants aged 12 to 24 months at enrollment; to receive Hepatitis A vaccine (Day 0) and Japanese encephalitis vaccine (Day 28)
  Interventions: Biological: Hepatitis A vaccine (Day 0) Japanese encephalitis vaccine (Day 28)

INTERVENTIONS:
Biological: Japanese encephalitis vaccine (Day 0) Hepatitis A vaccine (Day 28) — ≥4.0 Log10 Plaque forming units (PFU), Subcutaneous (SC; Day 0); 0.5 mL intramuscular (IM; Day 28)
  Other Names: ChimeriVax™-JE
  Arms: JE-CV/Hepatitis A (Group 1)
Biological: Hepatitis A vaccine (Day 0) Japanese encephalitis vaccine (Day 28) — 0.5 mL IM (Day 0); ≥4.0 Log10 PFU SC (Day 28)
  Other Names: ChimeriVax™-JE
  Arms: Hepatitis A/JE-CV (Group 2)
Biological: Japanese encephalitis vaccine (Day 0) Hepatitis A vaccine (Day 28) — ≥4.0 Log10 PFU SC (Day 0); 0.5 mL IM (Day 28)
  Other Names: ChimeriVax™-JE
  Arms: JE-CV/Hepatitis A (Group 3)
Biological: Hepatitis A vaccine (Day 0) Japanese encephalitis vaccine (Day 28) — 0.5 mL IM (Day 0); ≥4.0 Log10 PFU SC (Day 28)
  Other Names: ChimeriVax™-JE
  Arms: Hepatitis A/JE-CV (Group 4)

SUMMARY:
Safety:

To describe the safety profiles following vaccination.

Immunogenicity:

To describe the immune response after a single dose of vaccine.

DETAILED DESCRIPTION:
This is a randomized, cross-over, open, active controlled, multi-center trial in toddlers and children in Thailand. Stepwise enrollment of children in 2 age cohorts. Subjects will be followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of consent form signed by at least one parent or another legally acceptable representative, and by at least one independent witness.
* Completion of vaccinations according to the national immunization schedule
* Subject and parent/legally acceptable representative able to attend all scheduled visits and comply with all trial procedures.
* Previous receipt of two doses of a mouse-brain-derived JE vaccine at 12 to 15 months of age according to the national immunization schedule and aged 2 to 5 years on the day of inclusion.
* Aged 12 to 24 months on the day of inclusion and have not received any JE vaccine.

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances.
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of the immune response.
* Receipt of hepatitis A vaccine.
* History of flavivirus infection (confirmed either clinically, serologically or microbiologically).
* Administration of any anti-viral within 2 months preceding the screening visit.
* History of central nervous system disorder or disease.
* Personal or family history of thymic pathology (thymoma), thymectomy, or myasthenia.
* Planned participation in another clinical trial during the present trial period.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination.
* Personal human immunodeficiency virus, hepatitis B or hepatitis C seropositivity in the blood sample taken at screening.
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination.
* Previous vaccination against flavivirus disease at any time before the trial other than a mouse-brain-derived JE vaccine given in a two-dose regimen at 12 to 15 months of age in accordance with the national immunization schedule.
* Febrile illness or any acute illness/infection on the day of vaccination, according to investigator judgment
* History of seizures.
* Previous vaccination against flavivirus disease.

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Bangkok, Thailand

REFERENCES:
- [Result] Chokephaibulkit K, Sirivichayakul C, Thisyakorn U, Sabchareon A, Pancharoen C, Bouckenooghe A, Gailhardou S, Boaz M, Feroldi E. Safety and immunogenicity of a single administration of live-attenuated Japanese encephalitis vaccine in previously primed 2- to 5-year-olds and naive 12- to 24-month-olds: multicenter randomized controlled trial. Pediatr Infect Dis J. 2010 Dec;29(12):1111-7. doi: 10.1097/INF.0b013e3181f68e9c. PMID 20856164
- [Derived] Feroldi E, Boaz M, Yoksan S, Chokephaibulkit K, Thisyakorn U, Pancharoen C, Monfredo C, Bouckenooghe A. Persistence of Wild-Type Japanese Encephalitis Virus Strains Cross-Neutralization 5 Years After JE-CV Immunization. J Infect Dis. 2017 Jan 15;215(2):221-227. doi: 10.1093/infdis/jiw533. PMID 27815383
- [Derived] Chokephaibulkit K, Sirivichayakul C, Thisyakorn U, Pancharoen C, Boaz M, Bouckenooghe A, Feroldi E. Long-term follow-up of Japanese encephalitis chimeric virus vaccine: Immune responses in children. Vaccine. 2016 Nov 4;34(46):5664-5669. doi: 10.1016/j.vaccine.2016.09.018. Epub 2016 Sep 27. PMID 27686833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 02 March 2008 to 06 January 2009 at 3 clinic centers in Thailand.
Pre-assignment Details: A total of 300 participants who met all of the inclusion and none of the exclusion criteria were randomized and vaccinated in this study.
Groups:
- JE-CV/Hepatitis A (Group 1): Children aged 2 to 5 years of age received one dose of Japanese Encephalitis ChimeriVax™ (JE-CV) as first vaccination and one dose of Hepatitis A as second vaccination 28 days apart
- Hepatitis A/JE-CV (Group 2): Children aged 2 to 5 years of age received one dose of Hepatitis A as first vaccination and one dose of JE-CV as second vaccination 28 days apart
- JE-CV/Hepatitis A (Group 3): Toddlers aged 12 to 24 months of age received one dose of JE-CV as first vaccination and one dose of Hepatitis A as second vaccination 28 days apart
- Hepatitis A/JE-CV (Group 4): Toddlers aged 12 to 24 months of age received one dose of Hepatitis A as first vaccination and one dose of JE-CV as second vaccination 28 days apart
Period: Overall Study
Arm/Group | JE-CV/Hepatitis A (Group 1) | Hepatitis A/JE-CV (Group 2) | JE-CV/Hepatitis A (Group 3) | Hepatitis A/JE-CV (Group 4)
Started | 50 | 50 | 101 | 99
Completed | 50 | 50 | 101 | 98
Not Completed | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- JE CV/Hepatitis A (Group 1): Children aged 2 to 5 years of age received one dose of Japanese Encephalitis ChimeriVax™ (JE CV) as first vaccination and one dose of Hepatitis A as second vaccination 28 days apart
- Hepatitis A/JE CV (Group 2): Children aged 2 to 5 years of age received one dose of Hepatitis A as first vaccination and one dose of JE CV as second vaccination 28 days apart
- JE CV/Hepatitis A (Group 3): Toddlers aged 12 to 24 months of age received one dose of JE CV as first vaccination and one dose of Hepatitis A as second vaccination 28 days apart
- Hepatitis A/JE CV (Group 4): Toddlers aged 12 to 24 months of age received one dose of Hepatitis A as first vaccination and one dose of JE CV as second vaccination 28 days apart
- Total: Total of all reporting groups
Arm/Group | JE CV/Hepatitis A (Group 1) | Hepatitis A/JE CV (Group 2) | JE CV/Hepatitis A (Group 3) | Hepatitis A/JE CV (Group 4) | Total
Number analyzed (Participants) | 50 | 50 | 101 | 99 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 101 | 99 | 300
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 2.4 (0.5) | 2.5 (0.6) | 1.4 (0.2) | 1.3 (0.2) | 1.7 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 35 | 57 | 57 | 166
  Male | 33 | 15 | 44 | 42 | 134
Region of Enrollment [Number; unit: Participants]
  Thailand | 50 | 50 | 101 | 99 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Injection Site and Systemic Reactions After Injection With Either JE-CV or Hepatitis A Vaccine as First Injection
Description: 12 to 24 months - Injection site: Tenderness, Erythema, and Swelling; Systemic reactions: Fever, Vomiting, Crying Abnormal, Drowsiness, Appetite lost, and Irritability. Grade 3: Tenderness, Cries if limb is moved; Erythema and Swelling, ≥5 cm; Fever, >39.5˚C; Vomiting, ≥ 6 times/day; Abnormal crying, >3 hours; Drowsiness, Sleeping often; Appetite lost, Refuses ≥3 feeds/meals; Irritability, Inconsolable.
  2 to 5 years - Injection site: Pain, Erythema, and Swelling; Systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia. Grade 3: Pain, Incapacitating; Erythema and Swelling, ≥5 cm; Fever, >39˚C; Headache, Malaise, and Myalgia, Prevents activities.
Time Frame: Day 0 up to Day 14 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set, which includes all persons who received at least one dose of study vaccine.
Measure: Number; unit: Participants
Arm/Group | JE-CV/Hepatitis A (Group 1) | Hepatitis A/JE-CV (Group 2) | JE-CV/Hepatitis A (Group 3) | Hepatitis A/JE-CV (Group 4)
Number analyzed (Participants) | 50 | 50 | 101 | 99
Participants
  Injection site Pain (N=50,50,0,0) | 15 | 13 [0 to 0] | NA [0 to 0] — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group
  Grade 3 Injection site Pain (N=50,50,0,0) | 0 | 0 [0 to 0] | NA [0 to 0] — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group
  Injection site Tenderness (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 43 [0 to 0] | 19 [0 to 0]
  Grade 3 Injection site Tenderness (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 0 [0 to 0] | 0 [0 to 0]
  Injection site Erythema (N=50,50,101,99) | 7 | 9 [0 to 0] | 23 [0 to 0] | 16 [0 to 0]
  Grade 3 Injection site Erythema (N=50,50,101,99) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Injection site Swelling (N=50,50,101,99) | 4 | 5 [0 to 0] | 6 [0 to 0] | 8 [0 to 0]
  Grade 3 Swelling (N=50,50,101,99) | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Fever (N=50,50,101,99) | 8 | 8 [0 to 0] | 14 [0 to 0] | 18 [0 to 0]
  Grade 3 Fever (N=50,50,101,99) | 1 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Headache (N=50,50,0,0) | 7 | 7 [0 to 0] | NA [0 to 0] — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group
  Grade 3 Headache (N=50,50,0,0) | 0 | 0 [0 to 0] | NA [0 to 0] — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group
  Malaise (N=50,50,0,0) | 15 | 13 [0 to 0] | NA [0 to 0] — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group
  Grade 3 Malaise (N=50,50,0,0) | 0 | 0 [0 to 0] | NA [0 to 0] — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group
  Myalgia (N=50,50,0,0) | 14 | 8 [0 to 0] | NA [0 to 0] — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group
  Grade 3 Myalgia (N=50,50,0,0) | 0 | 0 [0 to 0] | NA [0 to 0] — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group
  Vomiting (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 21 [0 to 0] | 21 [0 to 0]
  Grade 3 Vomiting (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 1 [0 to 0] | 0 [0 to 0]
  Crying abnormal (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 24 [0 to 0] | 20 [0 to 0]
  Grade 3 Crying abnormal (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 0 [0 to 0] | 0 [0 to 0]
  Drowsiness (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 22 [0 to 0] | 13 [0 to 0]
  Grade 3 Drowsiness (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 0 [0 to 0] | 0 [0 to 0]
  Appetite lost (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 28 [0 to 0] | 32 [0 to 0]
  Grade 3 Appetite lost (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 0 [0 to 0] | 2 [0 to 0]
  Irritability (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 32 [0 to 0] | 24 [0 to 0]
  Grade 3 Irritability (N=0,0,101,99) | NA — This safety event was not solicited for this group | NA [0 to 0] — This safety event was not solicited for this group | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Number of Participants With Solicited Injection Site and Systemic Reactions After Injection With Either JE-CV or Hepatitis A Vaccine as Second Injection
Description: as for outcome 1
Time Frame: Day 0 up to Day 14 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set, which includes all persons who received at least one dose of study vaccine. A participant in Group 1 was given JE-CV vaccine as the second vaccination in error; and counted for Group 2 for the safety outcome for the second injection.
Measure: Number; unit: Participants
Arm/Group | JE-CV/Hepatitis A (Group 1) | Hepatitis A/JE-CV (Group 2) | JE-CV/Hepatitis A (Group 3) | Hepatitis A/JE-CV (Group 4)
Number analyzed (Participants) | 48 | 51 | 101 | 98
Participants
  Injection site Pain (N=48,51,0,0) | 15 | 9 | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group
  Grade 3 Injection site Pain (N=48,51,0,0) | 0 | 0 | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group
  Injection site Tenderness (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 35 | 20
  Grade 3 Injection site Tenderness (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 1 | 0
  Injection site Erythema (N=48,51,100,98) | 8 | 7 | 23 | 22
  Grade 3 Injection site Erythema (N=48,51,100,98) | 0 | 0 | 0 | 0
  Injection site Swelling (N=48,51,100,98) | 8 | 4 | 6 | 11
  Grade 3 Swelling (N=48,51,100,98) | 0 | 0 | 0 | 0
  Fever (N=48,51,100,98) | 5 | 14 | 23 | 28
  Grade 3 Fever (N=48,51,100,98) | 1 | 0 | 1 | 2
  Headache (N=48,51,0,0) | 7 | 14 | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group
  Grade 3 Headache (N=48,51,0,0) | 0 | 0 | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group
  Malaise (N=48,51,0,0) | 13 | 18 | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group
  Grade 3 Malaise (N=48,51,0,0) | 0 | 0 | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group
  Myalgia (N=48,51,0,0) | 7 | 10 | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group
  Grade 3 Myalgia (N=48,51,0,0) | 0 | 0 | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group
  Vomiting (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 23 | 19
  Grade 3 Vomiting (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 1 | 1
  Crying abnormal (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 19 | 21
  Grade 3 Crying abnormal (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 2 | 0
  Drowsiness (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 17 | 14
  Grade 3 Drowsiness (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 0 | 0
  Appetite lost (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 26 | 24
  Grade 3 Appetite lost (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 2 | 1
  Irritability (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 22 | 24
  Grade 3 Irritability (N=0,0,100,98) | NA — This safety event was not solicited for this group | NA — This safety event was not solicited for this group | 1 | 0

3. Secondary Outcome: Percentage of Participants With Seroconversion to JE-CV Vaccine Antigens Following Administration of JE-CV Vaccination
Description: JE virus neutralizing antibody measurement was assessed by plaque reduction neutralization test (PRNT50). Seroconversion was defined as participants with a pre-vaccination titer < 10 (1/dil) and post-vaccination titer ≥ 10 (1/dil), or participants with pre-vaccination titer ≥ 10 (1/dil) and 4-fold increase from pre- to post-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Seroconversion to the JE-CV vaccine antigens was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | JE-CV/Hepatitis A (Group 1) | Hepatitis A/JE-CV (Group 2) | JE-CV/Hepatitis A (Group 3) | Hepatitis A/JE-CV (Group 4)
Number analyzed (Participants) | 49 | 48 | 87 | 95
Percentage of participants
  Homologous virus (N=49,48,83,88) | 89.8 | 95.8 [0 to 0] | 100.0 [0 to 0] | 93.2 [0 to 0]
  Genotype I (N=49,48,81,91) | 83.7 | 93.8 [0 to 0] | 98.8 [0 to 0] | 95.6 [0 to 0]
  Genotype II (N=49,48,81,91) | 83.7 | 93.8 [0 to 0] | 96.3 [0 to 0] | 95.6 [0 to 0]
  Genotype III (N=49,48,81,93) | 87.8 | 91.7 [0 to 0] | 100.0 [0 to 0] | 94.6 [0 to 0]
  Genotype IV (N=49,48,81,90) | 89.8 | 91.7 [0 to 0] | 74.1 [0 to 0] | 65.6 [0 to 0]

4. Secondary Outcome: Summary of Geometric Mean Titers Against JE Antibodies Before and After JE-CV Vaccination
Description: JE virus neutralizing antibody measurement was assessed by the PRNT50 assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Geometric mean titers against the JE-CV vaccine antigens were assessed in the Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | JE-CV/Hepatitis A (Group 1) | Hepatitis A/JE-CV (Group 2) | JE-CV/Hepatitis A (Group 3) | Hepatitis A/JE-CV (Group 4)
Number analyzed (Participants) | 49 | 48 | 87 | 95
Titers
  Homologous virus (pre-vaccination; N=49,48,86,90) | 49.5 [33.9 to 72.1] | 40.6 [26.4 to 62.4] | 5.78 [5.25 to 6.37] | 5.08 [4.92 to 5.24]
  Homologous virus (post-vaccination; N=49,48,84,93) | 1957 [1227 to 3120] | 3568 [2361 to 5394] | 500 [353 to 708] | 167 [120 to 233]
  Genotype I (pre-vaccination; N=49,48,83,91) | 55.2 [36.0 to 84.6] | 55.3 [35.3 to 86.7] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Genotype I (post-vaccination; N=49,48,82,94) | 1016 [703 to 1467] | 1988 [1427 to 2770] | 170 [130 to 223] | 155 [117 to 206]
  Genotype II (pre-vaccination; N=49,48,83,91) | 46.5 [31.9 to 67.9] | 34.2 [22.7 to 51.4] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Genotype II (post-vaccination; N=49,48,82,94) | 921 [625 to 1356] | 1566 [1090 to 2250] | 157 [119 to 206] | 121 [93.7 to 156]
  Genotype III (pre-vaccination; N=49,48,83,93) | 39.2 [27.0 to 57.0] | 40.6 [25.7 to 64.0] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Genotype III (post-vaccination; N=49,48,82,94) | 1107 [726 to 1689] | 2089 [1405 to 3105] | 189 [140 to 255] | 98.2 [73.2 to 132]
  Genotype IV (pre-vaccination; N=49,48,83,90) | 25.2 [18.1 to 35.1] | 20.0 [13.8 to 28.9] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Genotype IV (post-vaccination; N=49,48,82,94) | 604 [387 to 944] | 829 [575 to 1195] | 25.3 [19.1 to 33.5] | 17.0 [13.6 to 21.3]

5. Other Pre Specified Outcome: Summary of Persistence of Seroprotection to JE-CV Antigens Up To Five Years Following Vaccination
Description: Japanese Encephalitis virus neutralizing antibody measurement was assessed by the PRNT50 assay.
Time Frame: Day 0 (pre-vaccination) up to 5 years after final vaccination
Population: Persistence of seroprotection to JE-CV antigens was assessed in the Full Analysis Set.
Measure: Number; unit: Participants
Arm/Group | JE-CV/Hepatitis A (Group 1) | Hepatitis A/JE-CV (Group 2) | JE-CV/Hepatitis A (Group 3) | Hepatitis A/JE-CV (Group 4)
Number analyzed (Participants) | 50 | 50 | 101 | 99
Participants
  Homologous virus (pre-vaccination; N=50,50,100,94) | 45 | 41 [0 to 0] | 15 [0 to 0] | 2 [0 to 0]
  Homologous virus (post-vaccination; N=49,50,98,96) | 49 | 50 [0 to 0] | 98 [0 to 0] | 89 [0 to 0]
  Homologous virus (post-6 months; N=48,49,99,98) | 48 | 49 [0 to 0] | 91 [0 to 0] | 80 [0 to 0]
  Homologous virus (post-1 year; N=48,45,91,89) | 46 | 44 [0 to 0] | 81 [0 to 0] | 71 [0 to 0]
  Homologous virus (post-2 years; N=43,41,85,79) | 41 | 41 [0 to 0] | 74 [0 to 0] | 64 [0 to 0]
  Homologous virus (post-3 years; N=40,38,68,56) | 40 | 38 [0 to 0] | 66 [0 to 0] | 52 [0 to 0]
  Homologous virus (post-4 years; N=41,36,63,56) | 41 | 36 [0 to 0] | 63 [0 to 0] | 54 [0 to 0]
  Homologous virus (post-5 years; N=40,38,60,50) | 40 | 38 [0 to 0] | 55 [0 to 0] | 44 [0 to 0]
  Genotype I (pre-vaccination; N=50,50,97,95) | 40 | 41 [0 to 0] | 8 [0 to 0] | 3 [0 to 0]
  Genotype I (post-vaccination; N=49,50,96,97) | 49 | 50 [0 to 0] | 95 [0 to 0] | 93 [0 to 0]
  Genotype I (post-6 months; N=47,48,99,98) | 47 | 48 [0 to 0] | 95 [0 to 0] | 86 [0 to 0]
  Genotype II (pre-vaccination; N=49,50,97,95) | 39 | 39 [0 to 0] | 9 [0 to 0] | 2 [0 to 0]
  Genotype II (post-vaccination; N=49,50,96,97) | 49 | 50 [0 to 0] | 93 [0 to 0] | 93 [0 to 0]
  Genotype II (post-6 months; N=47,48,99,98) | 47 | 48 [0 to 0] | 90 [0 to 0] | 80 [0 to 0]
  Genotype III (pre-vaccination; N=50,50,97,97) | 41 | 38 [0 to 0] | 5 [0 to 0] | 1 [0 to 0]
  Genotype III (post-vaccination; N=49,50,96,97) | 49 | 50 [0 to 0] | 96 [0 to 0] | 92 [0 to 0]
  Genotype III (post-6 months; N=48,48,99,98) | 48 | 48 [0 to 0] | 73 [0 to 0] | 62 [0 to 0]
  Genotype IV (pre-vaccination; N=49,50,97,94) | 39 | 32 [0 to 0] | 5 [0 to 0] | 0 [0 to 0]
  Genotype IV (post-vaccination; N=49,50,96,97) | 48 | 50 [0 to 0] | 73 [0 to 0] | 65 [0 to 0]
  Genotype IV (post-6 months; N=47,48,99,98) | 47 | 48 [0 to 0] | 68 [0 to 0] | 46 [0 to 0]

6. Other Pre Specified Outcome: Summary of Geometric Mean Titer Against JE Antibodies Up To Five Years Following Vaccination With JE-CV Vaccine
Description: Japanese Encephalitis virus neutralizing antibody measurement was assessed by the PRNT50 assay.
Time Frame: Day 0 (pre-vaccination) up to 5 years after final vaccination
Population: Geometric Mean Titers Against JE Antibodies were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | JE-CV/Hepatitis A (Group 1) | Hepatitis A/JE-CV (Group 2) | JE-CV/Hepatitis A (Group 3) | Hepatitis A/JE-CV (Group 4)
Number analyzed (Participants) | 50 | 50 | 101 | 99
Titers
  Homologous virus (pre-vaccination; N=50,50,100,94) | 48.6 [33.5 to 70.4] | 41.1 [27.2 to 62.2] | 6.11 [5.51 to 6.78] | 5.15 [4.94 to 5.37]
  Homologous virus (post-vaccination; N=49,50,98,96) | 1956.7 [1227.1 to 3120.0] | 3722.2 [2489.2 to 5565.9] | 517.6 [371.7 to 720.9] | 167.1 [120.2 to 232.2]
  Homologous virus (post-6 months; N=48,49,99,98) | 892.1 [566.1 to 1405.8] | 1244.3 [798.8 to 1938.3] | 96.6 [71.4 to 130.9] | 49.8 [36.8 to 67.4]
  Homologous virus (post-1 year; N=48,45,91,89) | 339 [216 to 531] | 621 [382 to 1009] | 78.8 [57.8 to 107] | 49.0 [34.9 to 68.6]
  Homologous virus (post-2 years; N=43,41,85,79) | 414 [246 to 698] | 662 [403 to 1088] | 94.2 [66.0 to 134] | 67.1 [46.3 to 97.3]
  Homologous virus (post-3 years; N=40,38,68,56) | 422 [273 to 654] | 505 [339 to 751] | 146 [102 to 208] | 90.5 [62.6 to 131]
  Homologous virus (post-4 years; N=41,36,63,56) | 360 [223 to 582] | 559 [306 to 1023] | 137 [100 to 188] | 110 [77.5 to 157]
  Homologous virus (post-5 years; N=40,38,60,50) | 222 [151 to 328] | 287 [183 to 449] | 68.8 [48.3 to 98.1] | 58.2 [36.4 to 93.0]
  Genotype I (pre-vaccination; N=50,50,97,95) | 54.8 [36.1 to 83.3] | 55.3 [35.2 to 86.9] | 5.62 [5.18 to 6.11] | 5.18 [4.96 to 5.41]
  Genotype I (post-vaccination; N=49,50,96,97) | 1015.8 [703.4 to 1466.9] | 2116.7 [1519.8 to 2948.1] | 186.8 [142.2 to 245.3] | 163.1 [122.5 to 217.1]
  Genotype I (6-months; N=47,48,99,98) | 863.5 [573.9 to 1299.3] | 981.0 [678.4 to 1418.4] | 81.4 [62.8 to 105.5] | 52.4 [40.2 to 68.2]
  Genotype II (pre-vaccination; N=49,50,97,95) | 46.5 [31.9 to 67.9] | 33.3 [22.3 to 49.6] | 5.75 [5.16 to 6.40] | 5.20 [4.90 to 5.53]
  Genotype II (post-vaccination; N=49,50,96,97) | 920.6 [624.9 to 1356.2] | 1763.4 [1199.3 to 2592.9] | 163.2 [125.5 to 212.3] | 126.8 [97.8 to 164.4]
  Genotype II (post-6 months; N=47,48,99,98) | 581.2 [402.9 to 838.3] | 714.4 [520.4 to 980.7] | 72.3 [54.4 to 96.1] | 42.4 [31.7 to 56.8]
  Genotype III (pre-vaccination; N=50,50,97,97) | 37.6 [25.8 to 54.7] | 41.1 [26.5 to 63.7] | 5.39 [5.04 to 5.76] | 5.08 [4.93 to 5.23]
  Genotype III (post-vaccination; N=49,50,96,97) | 1107.1 [725.8 to 1688.7] | 2210.4 [1498.2 to 3261.0] | 200.2 [151.5 to 264.6] | 102.1 [75.8 to 137.6]
  Genotype III (post-6 months; N=48,48,99,98) | 513.1 [326.5 to 806.5] | 645.7 [438.7 to 950.4] | 31.1 [23.3 to 41.5] | 20.2 [15.6 to 26.3]
  Genotype IV (pre-vaccination; N=49,50,97,94) | 25.2 [18.1 to 35.1] | 19.7 [13.8 to 28.2] | 5.31 [5.03 to 5.60] | 5.00 [5.00 to 5.00]
  Genotype IV (post-vaccination; N=49,50,96,97) | 604.0 [386.6 to 943.6] | 874.0 [610.0 to 1252.3] | 28.5 [21.5 to 37.7] | 18.1 [14.3 to 23.0]
  Genotype IV (post-6 months; N=47,48,99,98) | 279.4 [194.1 to 402.3] | 363.4 [256.8 to 514.3] | 21.0 [16.2 to 27.2] | 12.6 [9.93 to 16.0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination.
Arm/Group | JE CV/Hepatitis A (Group 1) | Hepatitis A/JE CV (Group 2) | JE CV/Hepatitis A (Group 3) | Hepatitis A/JE CV (Group 4)
Serious Adverse Events (participants affected / at risk) | 3/50 | 3/50 | 11/101 | 10/99
Other Adverse Events (participants affected / at risk) | 15/50 | 18/50 | 43/101 | 35/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JE CV/Hepatitis A (Group 1) (N=50) | Hepatitis A/JE CV (Group 2) (N=50) | JE CV/Hepatitis A (Group 3) (N=101) | Hepatitis A/JE CV (Group 4) (N=99)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | JE CV/Hepatitis A (Group 1) (N=50) | Hepatitis A/JE CV (Group 2) (N=50) | JE CV/Hepatitis A (Group 3) (N=101) | Hepatitis A/JE CV (Group 4) (N=99)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3/48 (3) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5) | 5 (5) | 11 (12)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 8 (8) | 35 (35) | 35 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 13 (16) | 11 (12)
Heat rash (Skin and subcutaneous tissue disorders) | 3/48 (4) | 0 (0) | 0 (0) | 0 (0)
Injection-site pain (General disorders) | 15/48 (15) | 13 (13) | 0/0 (0) | 0/0 (0)
Injection-site tenderness (General disorders) | 0/0 (0) | 0/0 (0) | 43 (43) | 20/98 (20)
Injection-site erythema (General disorders) | 8/48 (8) | 9 (9) | 23/100 (23) | 22/98 (22)
Injection-site swelling (General disorders) | 8/48 (8) | 5 (5) | 6/100 (6) | 11/98 (11)
Fever (General disorders) | 8 (8) | 14 (14) | 23/100 (23) | 28/98 (28)
Headache (Nervous system disorders) | 7/48 (7) | 14 (14) | 0/0 (0) | 0/0 (0)
Malaise (General disorders) | 15 (15) | 18 (18) | 0/0 (0) | 0/0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 10 (10) | 0/0 (0) | 0/0 (0)
Vomiting (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 23/100 (23) | 21 (21)
Crying abnormal (Psychiatric disorders) | 0/0 (0) | 0/0 (0) | 24 (24) | 21/98 (21)
Drowsiness (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 22 (22) | 14/98 (14)
Appetite lost (Metabolism and nutrition disorders) | 0/0 (0) | 0/0 (0) | 28 (28) | 32 (32)
Irritability (Psychiatric disorders) | 0/0 (0) | 0/0 (0) | 32 (32) | 24/98 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.